CLINICAL TRIAL: NCT02845037
Title: A Rising Single Oral Dose Study to Investigate the Tolerability, Pharmacokinetics and Dopamine ß-hydroxylase (DßH) Inhibition Profile of BIA 5-453 in Healthy Male Volunteers
Brief Title: Tolerability, Pharmacokinetics and Dopamine ß-hydroxylase (DßH) Inhibition Profile of BIA 5-453
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-5453-101
Record Dates: First submitted 2016-07-15; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Chronic Heart Failure
MeSH Terms: conditions — Hypertension | interventions — etamicastat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 2 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 10 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 20 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 50 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 100 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 200 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 400 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 600 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 900 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo
- 1200 mg or placebo (Experimental): BIA 5-453 or placebo
  Interventions: Drug: BIA 5-453; Drug: Placebo

INTERVENTIONS:
Drug: BIA 5-453 — BIA 5-453 Gelatine capsule for oral administration (1, 10 or 20 mg). Single oral doses of BIA 4-543 2 mg, 10 mg, 20 mg, 50 mg, 100 mg, 200 mg, 400 mg, 600 mg, 900 mg and 1200 mg were administered to subjects in fasting conditions.
  Other Names: Etamicastat
Drug: Placebo — Placebo Gelatine capsule for oral administration. The composition of the placebo is qualitatively the same but without BIA 5-453 pharmaceutical active ingredient (API).
  Other Names: Placebo Gelatine capsule

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BIA 5-453 after single oral doses

DETAILED DESCRIPTION:
Single centre, randomised, double-blind, placebo-controlled study of single ascending doses in 10 sequential groups of 8 healthy young male volunteers. Within each group (n=8), 6 volunteers were randomised to receive BIA 5-453 and the remaining 2 volunteers were randomised to receive placebo. A volunteer participated only in a single period.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated informed consent form before any study-specific screening procedure was performed.
2. Aged between 18 and 45 years, inclusive.
3. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12-lead electrocardiogram (ECG).
4. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must have been able to abstain from smoking during the inpatient stay.
5. Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

Medical History

1. Any significant cardiovascular (e.g. hypertension), hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunologic, dermatological, haematological, neurologic, or psychiatric disease.
2. Acute disease state (e.g., nausea, vomiting, fever, diarrhoea) within 7 days before study day 1.
3. History of drug abuse within 1 year before study day 1.
4. History of alcoholism within 1 year before day 1. Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g
5. History of any clinically important drug allergy.

   Physical and Laboratory Findings
6. An automatic ECG QTc interval reading at screening or enrolment >450 ms.
7. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
8. Positive findings of urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA [3,4-methylenedioxy-methamphetamine; ecstasy]).

   Prohibited treatments
9. Prohibited Treatments: use of any investigational drug within 90 days or prescription drug within 30 days before investigational medical product (IMP) administration.
10. Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 72 before study day -1.
11. Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before IMP administration.
12. Donation of blood (ie 450 ml) within 90 days before study day 1.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1 pre-dose then at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60, and 72 hours post-dose
  Mean BIA 5-453 plasma pharmacokinetic parameters ± SD following single doses of 2, 10, 20, 50, 100, 200, 400, 600, 900 and 1200 mg of BIA 5-453 in 10 groups of 6 healthy volunteers each
Time to reach Cmax (Tmax) | Day 1 pre-dose then at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60, and 72 hours post-dose
  Mean BIA 5-453 plasma pharmacokinetic parameters ± SD following single doses of 2, 10, 20, 50, 100, 200, 400, 600, 900 and 1200 mg of BIA 5-453 in 10 groups of 6 healthy volunteers each
Area under the plasma concentration-time curve from time 0 to the time of last quantifiable concentration (AUC0-t) | Day 1 pre-dose then at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60, and 72 hours post-dose
  Mean BIA 5-453 plasma pharmacokinetic parameters ± SD following single doses of 2, 10, 20, 50, 100, 200, 400, 600, 900 and 1200 mg of BIA 5-453 in 10 groups of 6 healthy volunteers each
Area under the plasma concentration-time curve from time 0 to the infinity (AUC0-∞) | Day 1 pre-dose then at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60, and 72 hours post-dose
  Mean BIA 5-453 plasma pharmacokinetic parameters ± SD following single doses of 2, 10, 20, 50, 100, 200, 400, 600, 900 and 1200 mg of BIA 5-453 in 10 groups of 6 healthy volunteers each
% of subjects with at least one adverse event | through study completion, an average of 72 hours
  Adverse events were continuously monitored from screening until the follow-up visit.
% of subjects by dose group with at least one treatment-emergent adverse event (TEAEs) | through study completion, an average of 72 hours
  Treatment emergent adverse events (TEAE) were defined as adverse events which did not exist before dosing and appeared in the 72 hours following treatment administration or which was present before administration and worsened in the 72 hours following treatment administration.
Apparent terminal elimination half-life (t1/2) | Day 1 pre-dose then at 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, 48, 60, and 72 hours post-dose
  Mean BIA 5-453 plasma pharmacokinetic parameters ± SD following single doses of 2, 10, 20, 50, 100, 200, 400, 600, 900 and 1200 mg of BIA 5-453 in 10 groups of 6 healthy volunteers each

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided